CLINICAL TRIAL: NCT04632927
Title: A 28-week, Randomized, Double-blind, Active Controlled, Multicenter Study to Evaluate the Efficacy of Subcutaneously Administered Secukinumab Compared to Ustekinumab in Adult Patients With Psoriatic Arthritis and Failure of TNFα- Inhibitor Treatment (AgAIN)
Brief Title: Efficacy of Secukinumab Compared to Ustekinumab in Adults With Active Psoriatic Arthritis and Failure of TNFα-Inhibitor Treatment
Acronym: AgAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457FDE04; 2019-004246-15 (EudraCT Number)
Record Dates: First submitted 2020-11-04; First posted 2020-11-17 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Psoriasis Arthropathica; Psoriatic Arthropathy
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): AIN457
  Interventions: Biological: Secukinumab; Biological: Ustekinumab
- Ustekinumab (Experimental)
  Interventions: Biological: Secukinumab; Biological: Ustekinumab

INTERVENTIONS:
Biological: Secukinumab — Eligible subjects are randomized to one of two treatment arms in a 1:1 ratio
  Other Names: AIN457
Biological: Ustekinumab — Eligible subjects are randomized to one of two treatment arms in a 1:1 ratio

SUMMARY:
The purpose of this study is to compare the safety and efficacy of secukinumab and ustekinumab in patients with active psoriatic arthritis who showed failure to previous TNFα-inhibitor treatment

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of PsA as classified by CASPAR criteria for at least 6 months before randomization.
* Active PsA at baseline defined as ≥ 3 tender joints out of 68 and ≥ 3 swollen joints out of 66 (dactylitis of a digit counts as one joint each).
* Inadequate response or intolerance to previous or current treatment with at least one TNFα inhibitor
* Inadequate response or intolerance to conventional disease modifying anti-rheumatic drugs (cDMARDs)
* Diagnosis of active plaque psoriasis, with at least one psoriatic plaque of ≥ 2 cm diameter and/or nail changes consistent with psoriasis and/or documented history of plaque psoriasis.
* Rheumatoid factor (RF) and anti-cyclic citrullinated peptide (CCP) antibodies negative at screening.

Key Exclusion Criteria:

* Pregnant or nursing women,
* Previous exposure to secukinumab, ustekinumab or any other biologic drug directly targeting IL-17, IL-17 receptor, IL-12 or IL-23.
* Patients for whom the use of secukinumab or ustekinumab is contraindicated.
* Use of any other investigational drug. Previous treatment with any cell-depleting therapies including but not limited to anti-CD20 or investigational agents
* Evidence of ongoing infectious or malignant process
* Subjects receiving high potency opioid analgesics
* Ongoing use of prohibited psoriasis treatments/medications

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Germany (23):
  - Novartis Investigative Site, Rendsburg, Schleswig-Holstein
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Ehringshausen
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gommern
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Planegg
  - Novartis Investigative Site, Ratingen

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized in 28 study sites across Germany
Pre-assignment Details: A total of 144 patients overall were screened and 25 patients failed screening, while 119 patients completed the screening period successfully and underwent randomization
Groups:
- Secukinumab: Participants received 300 mg of secukinumab, administered as two 150 mg subcutaneous (s.c.) injections. Treatment was administered in a double-blind manner at Baseline and at Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24.
- Ustekinumab: Participants received ustekinumab via s.c. injection containing 45 mg (for participants weighing ≤100 kg) or 90 mg (for participants >100 kg). One active injection was administered at Baseline, Week 4, and 16.
  To maintain the blind, secukinumab-matching placebo injections were administered at all treatment time points (Baseline and at Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24). Depending on whether an ustekinumab injection was scheduled, participants received either one or two placebo injections per time point.
Period: Overall Study
Arm/Group | Secukinumab | Ustekinumab
Started | 56 | 63
Completed | 56 | 53
Not Completed | 0 | 10
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 4
Not completed — Loss of efficacy | 0 | 1
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Subject decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Ustekinumab | Total
Number analyzed (Participants) | 56 | 63 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (8.8) | 52.7 (12.7) | 53.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 80
  Male | 17 | 22 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 55 | 62 | 117
  Black | 1 | 0 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Health Assessment Questionnaire - Disability Index (HAQ-DI) Response at Week 28
Description: The disability assessment component of the HAQ evaluated a subject's level of functional ability through 20 questions grouped into 8 categories: dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Each item began with the prompt "Over the past week, are you able to…" and is scored on a 4-point scale: 0 (no difficulty), 1 (some difficulty), 2 (much difficulty), and 3 (unable to do). The overall score was calculated by averaging the scores across all answered domains, resulting in a total score ranging from 0 (no disability) to 3 (severe disability).
  A HAQ-DI response was defined as an improvement of ≥0.35 points from baseline at Week 28. Missing values were imputed as non-responders
Time Frame: Baseline, Week 28
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment (investigational or control treatment) was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 63
Participants | 32 | 17
Statistical Analysis 1: Comparison: Secukinumab vs Ustekinumab; Test type: Other; p = 0.002, Regression, Logistic; The OR was calculated using a logistic regression model with treatment group, baseline HAQ-DI and strata (body weight) as independent variables; Odds Ratio (OR) = 3.647, 95% CI 2-sided [1.601 to 8.311]

2. Secondary Outcome: Number of Participants Achieving Psoriasis Area and Severity Index (PASI) 90 Response at Week 28
Description: The Psoriasis Area and Severity Index (PASI) was a composite measure that evaluates the average severity of erythema, induration, and desquamation of psoriatic lesions-each graded on a scale from 0 (none) to 4 (severe)-across four body regions: head, upper limbs, trunk (including groin), and lower limbs (to the top of the buttocks). These scores were weighted by the area of skin involvement in each region to generate a total PASI score ranging from 0 to 72, with higher scores indicating more severe disease activity.
  The number of participants who achieved at least a 90% reduction in PASI score from baseline at Week 28 was assessed. Missing values were imputed as non-responders.
Time Frame: Baseline, Week 28
Population: FAS: all patients to whom study treatment (investigational or control treatment) was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 63
Participants | 27 | 25

3. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain on VAS at Week 28
Description: The patient's level of pain was evaluated using a horizontal Visual Analogue Scale (VAS), on which individuals marked their pain intensity with a vertical tick. The scale ranged from 0 mm (indicating "no pain") to 100 mm (indicating "unbearable pain").
  The change in the patient's pain assessment on the VAS from baseline to Week 28 was analyzed. A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 28
Population: FAS: all patients to whom study treatment (investigational or control treatment) was assigned by randomization.
  Only participants with both a baseline and a Week 28 assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 58
Score on a Scale | -27.1 (25.8) | -16.4 (24.2)

4. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) 68 at Week 28
Description: Tender joint count (TJC) 68 was a method of assessing joint inflammation. Number of tender joints was determined by examining 68 joints and identifying the joints that were painful under pressure or to passive motion. The 68 joints assessed for tenderness included the 2 temporomandibular, 2 sternoclavicular, 2 acromioclavicular joints, 2 shoulders, 2 elbows, 2 wrists, 10 metacarpophalangeal, 10 proximal interphalangeal, 8 distal interphalangeal joints of the hands, 2 hips, 2 knees, 2 talo¬tibial, 2 mid-tarsal, 10 metatarsophalangeal, and 10 proximal interphalangeal joints of the feet.
  The change from baseline in TJC68 at Week 28 was assessed. A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 59
Score on a Scale | -9.6 (11.9) | -7.6 (10.7)

5. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) 66 at Week 28
Description: Swollen Joint Count (SJC) 66 was a method of assessing joint inflammation. The number of swollen joints was determined by examining 66 joints and identifying those with visible or palpable swelling suggestive of synovitis. The 66 joints assessed for swelling included the 2 sternoclavicular, 2 acromioclavicular joints, 2 shoulders, 2 elbows, 2 wrists, 10 metacarpophalangeal, 10 proximal interphalangeal, 8 distal interphalangeal joints of the hands, 2 knees, 2 talotibial, 2 mid-tarsal, 10 metatarsophalangeal, and 10 proximal interphalangeal joints of the feet.
  The change from baseline in SJC66 at Week 28 was assessed. A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 59
Score on a Scale | -6.8 (6.3) | -5.3 (5.2)

6. Secondary Outcome: Number of Patients Achieving PASI 100 at Week 28
Description: The PASI was a composite measure that evaluates the average severity of erythema, induration, and desquamation of psoriatic lesions-each graded on a scale from 0 (none) to 4 (severe)-across four body regions: head, upper limbs, trunk (including groin), and lower limbs (to the top of the buttocks). These scores were weighted by the area of skin involvement in each region to generate a total PASI score ranging from 0 to 72, with higher scores indicating more severe disease activity.
  The number of participants who achieved 100% reduction in PASI score from baseline at Week 28 was assessed. Missing values were imputed as non-responders.
Time Frame: Bseline, Week 28
Population: FAS: all patients to whom study treatment (investigational or control treatment) was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 63
Participants | 21 | 17

7. Secondary Outcome: Number of Patients Achieving PASI 75 at Week 28
Description: The Psoriasis Area and Severity Index (PASI) was a composite measure that evaluates the average severity of erythema, induration, and desquamation of psoriatic lesions-each graded on a scale from 0 (none) to 4 (severe)-across four body regions: head, upper limbs, trunk (including groin), and lower limbs (to the top of the buttocks). These scores were weighted by the area of skin involvement in each region to generate a total PASI score ranging from 0 to 72, with higher scores indicating more severe disease activity.
  The number of participants who achieved at least a 75% reduction in PASI score from baseline at Week 28 was assessed. Missing values were imputed as non-responders.
Time Frame: Baseline, Week 28
Population: FAS: all patients to whom study treatment (investigational or control treatment) was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 63
Participants | 34 | 29

8. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity on VAS
Description: The patient's global assessment of disease activity was performed using a 100 mm (VAS) ranging from 0 (='very good') to 100 (='very poor') after the question 'Considering all the ways Psoriatic Arthritis affects you, please indicate with a vertical mark through the horizontal line how well you are today'.
  The change in the patient's global assessment on the VAS from baseline to Week 28 was analyzed. A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 57
Score on a Scale | -26.0 (21.8) | -15.5 (23.1)

9. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Psoriasis and Arthritis Disease Activity on VAS
Description: The patient's assessment of psoriasis and arthritis was performed using a 100 mm VAS ranging from 0 (='Excellent') to 100 (='Poor') after the question 'Considering all the ways PSORIASIS and ARTHRITIS affects you, please indicate with a vertical mark through the horizontal line how well you are doing over the past week'
  The change in the patient's global assessment of psoriasis and arthritis disease activity on the VAS from baseline to Week 28 was analyzed. A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 58
Score on a Scale | -28.1 (23.6) | -16.2 (24.8)

10. Secondary Outcome: Number of Patients Achieving Minimal Disease Activity (MDA) at Week 28
Description: MDA was a composite endpoint used to assess low disease activity in patients with psoriatic arthritis and psoriasis. A patient was considered to have achieved MDA if they met at least 5 of the following 7 criteria:
  * TJC (0-68)≤1
  * SJC (0-66 joints)≤1
  * PASI ≤1 [the total score ranged from 0 (no disease) to 72 (maximal disease)] or body surface area≤3%
  * Patient's pain VAS ≤ 15 mm on a 100 mm scale, where 0 ="no pain" and 100= "pain as severe as can be imagined"
  * Patient's global assessment of disease activity (PtGA) ≤ 20 mm on a 100 mm scale, where 0 represented the lowest level of disease activity and 100 the highest
  * HAQ-DI ≤ 0.5, where 0 represented no difficulty and 3 represented inability to perform activities
  * Enthesitis count ≤ 1, based on the Leeds Enthesitis Index, where 0 indicated no tenderness and 6 indicated tenderness at all assessed tendon insertions
  The number of participants achieving MDA at Week 28 was assessed. Missing values were imputed as non-responders.
Time Frame: Week 28
Population: FAS: all patients to whom study treatment (investigational or control treatment) was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 63
Participants | 20 | 14

11. Secondary Outcome: Change From Baseline in the Leeds Enthesitis Index (LEI)
Description: The LEI was a validated enthesitis index that used six sites to evaluate enthesitis: the left and right lateral epicondyles of the humerus, the left and right proximal Achilles tendon insertions, and the left and right medial femoral condyles.Each site was scored as 0 (non-tender) or 1 (tender), resulting in a total score ranging from 0 to 6. A higher score reflected a greater burden of enthesitis.
  The change in the LEI score from baseline to Week 28 was analyzed. A negative change from baseline indicated an improvement in enthesitis severity
Time Frame: Baseline, Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 59
Score on a Scale | -0.9 (1.8) | -0.5 (1.5)

12. Secondary Outcome: Change From Baseline in the Leeds Dactylitis Index (LDI)
Description: The LDI was used to quantitatively assess dactylitis by measuring the circumference of affected digits and their corresponding control digits, along with the tenderness of each affected digit. Digits were classified as dactylitic if there was a ≥10% difference in circumference compared to the contralateral digit. When both digits were affected or a contralateral control was unavailable, a standardized reference range was applied.
  For each dactylitic digit, the ratio of the affected to control circumference was multiplied by a binary tenderness score (1 = tender, 0 = non-tender). The resulting values were summed across all affected digits to calculate the total LDI score. Scores ranged from 0 to 20, with higher scores indicating more severe or widespread dactylitis.
  The change in the LDI score from baseline to Week 28 was analyzed. A negative change from baseline indicated an improvement in dactylitis severity.
Time Frame: Baseline, Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 59
Score on a Scale | -9.7 (27.2) | -7.2 (25.9)

13. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Quality of Life (PsAQoL)
Description: The PsAQoL questionnaire was used to assess the impact of psoriatic arthritis on patients' quality of life. The PsAQoL is a validated, disease-specific, self-administered instrument consisting of 20 items with binary response options ("true" or "not true"). Items covered physical, emotional, and social domains, including fatigue, independence, and interpersonal relationships. The total score ranged from 0 to 20, with higher scores indicating greater impairment in quality of life.
  The change in the PsAQoL score from baseline to Week 28 was analyzed. A negative change from baseline indicated an improvement in health-related quality of life.
Time Frame: Baseline, Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 42 | 51
Score on a Scale | -2.5 (5.1) | -2.0 (5.4)

14. Secondary Outcome: Percentage of Participants Achieving a Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Response at Week 28
Description: The FACIT-Fatigue Scale was used to assess fatigue and its impact on daily functioning over the previous 7 days. The instrument consisted of 13 self-administered items, each scored on a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("Very much"). The total score ranged from 0 to 52, with higher scores indicating less fatigue and better functioning.
  Response was achieved if the score had improved by at least 4 points from baseline. Missing values were imputed as non-responders
Time Frame: Baseline, Week 28
Population: FAS: all patients to whom study treatment (investigational or control treatment) was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 63
Participants | 40 | 32

15. Secondary Outcome: Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) Response at Week 28
Description: The DLQI was used to evaluate the impact of dermatological conditions on patients' quality of life over the previous 7 days. It consisted of 10 self-administered items covering symptoms, daily activities, leisure, work/school, personal relationships, and treatment burden. Each item was scored from 0 ("Not at all") to 3 ("Very much"), with a total score ranging from 0 to 30. Higher scores indicated greater impairment.
  Response was achieved if the absolute score was either 0 or 1. Missing values were imputed as non-responders.
Time Frame: Week 28
Population: FAS: all patients to whom study treatment (investigational or control treatment) was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Ustekinumab
Number analyzed (Participants) | 56 | 63
Participants | 30 | 32

ADVERSE EVENTS:
Time Frame: From start of treatment to end of study, assessed up to approximately 36 weeks
Description: The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Groups:
- Secukinumab- On-Treatment; Ustekinumab - On-Treatment: AEs from start of treatment to 30 days after the last dose of study treatment, assessed up to approximately 28 weeks
- Secukinumab - Entire Study; Ustekinumab - Entire Study: AEs from start of treatment to end of study, assessed up to approximately 36 weeks
Arm/Group | Secukinumab- On-Treatment | Ustekinumab - On-Treatment | Secukinumab - Entire Study | Ustekinumab - Entire Study
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/63 | 0/56 | 0/63
Serious Adverse Events (participants affected / at risk) | 3/56 | 1/63 | 4/56 | 2/63
Other Adverse Events (participants affected / at risk) | 27/56 | 31/63 | 31/56 | 32/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab- On-Treatment (N=56) | Ustekinumab - On-Treatment (N=63) | Secukinumab - Entire Study (N=56) | Ustekinumab - Entire Study (N=63)
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Vertebrobasilar stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab- On-Treatment (N=56) | Ustekinumab - On-Treatment (N=63) | Secukinumab - Entire Study (N=56) | Ustekinumab - Entire Study (N=63)
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 5 | 4
COVID-19 (Infections and infestations) | 6 | 7 | 6 | 8
Nasopharyngitis (Infections and infestations) | 5 | 9 | 7 | 9
Respiratory tract infection (Infections and infestations) | 3 | 1 | 3 | 1
Urinary tract infection (Infections and infestations) | 4 | 5 | 5 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 3
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 6
Headache (Nervous system disorders) | 3 | 2 | 3 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 1 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT04632927/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT04632927/SAP_001.pdf